CLINICAL TRIAL: NCT00870129
Title: Using Advanced MR Imaging to Determine High Risk Areas in Patients With Malignant Gliomas and to Design Potential Radiation Plans: A Pilot Study, and to Examine Metabolite Changes in Gliomas and Other Solid Tumors
Brief Title: Magnetic Resonance (MR) Imaging to Determine High Risk Areas in Patients With Malignant Gliomas and to Design Potential Radiation Plans and to Examine Metabolite Changes in Gliomas and Other Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-009
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Brain Cancer; Glioma
Keywords: brain tumor; radiation; MRI; 09-009
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Magnetic Resonance Spectroscopy

ARMS (1):
- MRI (Experimental): The advanced MRI studies will be obtained at the time of the routinely scheduled preoperative planning MRI and/or the routinely scheduled pre-RT planning MRI at approximately 3±2 weeks after surgery. The routine sequences obtained for the planning MRI are standard of care. The advanced MRI sequences may or may not be additional as some have already been adopted into the standard of care imaging at MSKCC.
  Interventions: Procedure: MRI and advanced MRI sequences

INTERVENTIONS:
Procedure: MRI and advanced MRI sequences — This is a nonrandomized study in which each patient will receive the standard clinical care (in the form of surgery, radiation therapy and/or chemotherapy), as per the treating physician. Surgical resection will be performed at the discretion of the treating Neurooncologist and/or Neurooncology Tumor Board. Advanced brain MRIs with the 2 (or, in some cases, 3) special sequences will be obtained at the time of the clinically scheduled contrast MRIs, which are usually obtained immediately prior to and 1 months±3 weeks after radiation therapy if the patient requires radiation therapy for his/her tumor. The advanced brain MRI may also be obtained before surgery for suspected or confirmed gliomas, as per the standard of care, in some patients who may or may not require radiation therapy.

SUMMARY:
The researchers think that the use of advanced MR imaging may help people with this disease, because it may better predict areas within a malignant glioma (brain tumor) that are at a high risk of recurring. WeThe reserchers are doing this study to see whether this advanced imaging is a safe treatment that causes few or mild side effects in people with brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or Histopathologically proven diagnosis of high grade or low glioma or tumor is suspected to harbor an isocitrate dehydrogenase (IDH) mutation
* May undergo radiation therapy
* Patient and/or guardian is able to provide written informed consent prior to study registration
* Age ≥ 18 years old

Exclusion Criteria:

* Extreme claustrophobia that precludes MRI scan
* Known allergic reaction to Gd-DTPA
* Any contraindication to gadolinium intravenous contrast as per standard Department of Radiology contrast guidelines
* Any absolute contraindication to MRI (e.g., pacemaker, aneurysm clip, tissue expander).
* Pregnant or nursing female
* Unable to cooperate for MRI and/or radiation therapy planning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2009-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To assess the utility of baseline advanced MRI & changes between baseline & follow up advanced MRI in predicting high risk areas that are likely to develop progressive glioma despite chemoradiotherapy. | 1 -7 weeks before radiation treatment, about two months after treatment, and about every two months thereafter for the duration of the study.

SECONDARY OUTCOMES:
To compare radiation therapy simulations in patients with gliomas using conventional and baseline advanced MRI data. | prior to and 1 months±3 weeks after radiation therapy.
feasibility of 2HG spectroscopy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Young, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org